CLINICAL TRIAL: NCT06624553
Title: Effect of Monitoring With Freestyle Libre 2 Glucose Sensor on Treatment Satisfaction in Patients With Type 2 Diabetes Mellitus: Exploratory Study in Patients Starting Monitoring
Brief Title: Satisfaction With FreeStyle Libre 2 Monitoring Versus Capillary Blood Glucose Monitoring in People With DM2
Acronym: Diabetes type2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IIBSP-FSL-2021-150
Record Dates: First submitted 2024-08-07; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; glucose monitoring; satisfaction; diabetes technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Open and exploratory parallel randomized single-center clinical trial in a 1:1 ratio of three months duration. A computerized randomization by blocks of 10 without blinding will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group. Capilary glucose monitoring (No Intervention): The patient randomized to the control group, capillary glucose monitoring, will be provided with the necessary material for six weeks (Free Style Optium glucometer, puncturer, Free Style Optium strips, lancets and record book) and the objectives, technique of analysis, recording and interpretation. The patient/carer will be asked to practice before leaving the office to ensure that they perform the technique correctly and effectively.
- Intervention group. FreeStyle Libre 2 (Experimental): The patient randomized to the intervention group (FSL2) will be provided with the necessary material for six weeks (sensor, applicator and reader or mobile application (App)) and the objectives, analysis, recording and interpretation technique will be explained. The patient will be helped to register in the application and share the data with the hospital. The patient will carry out the first readings before leaving the consultation to ensure that they are carried out correctly.
  Interventions: Device: FreeStyle Libre 2, flash glucose monitoring

INTERVENTIONS:
Device: FreeStyle Libre 2, flash glucose monitoring — Currently, at the Hospital de la Santa Creu i Sant Pau, when starting monitoring in people with DM2, capillary glycemia monitoring is used, following the therapeutic education protocols in basal insulinization in the debut of DM2 and in optimization of treatment, protocols that are also applied to similar cases.
  The intervention group (FreeStyle Libre 2) will be provided with the necessary material to carry out the monitoring via a glucose sensor. Satisfaction with treatment will be assessed at the final study visit.
  Arms: Intervention group. FreeStyle Libre 2

SUMMARY:
The FreeStyle Libre 2 system is a Flash glucose monitoring system that, after a scan, provides information on interstitial glucose for the last 8 hours in the form of a reading every 15 min. The system is approved for non-adjuvant use for therapeutic decision-making. The acceptability and effectiveness of the FSL is well documented in patients with type 1 and 2 diabetes mellitus (DM2). Most of the studies in patients with DM2 have been developed in patients with insulin treatment, either basal or with multiple doses.

For all these reasons, we proposed an exploratory study to evaluate satisfaction with treatment (main variable) in people with DM2 who start glucose monitoring in the Endocrinology Day Hospital context compared to patients who use capillary blood glucose monitoring. These are patients treated in a context of debut/acute decompensation/intercurrent pathology, who will not necessarily be using insulin treatment. The aim is to know if the use of FSL2 provides benefits of user satisfaction with the treatment, assessed with the Diabetes Treatment Satisfaction Questionnaire at the end of follow-up (mean score of all items); in this context.

DETAILED DESCRIPTION:
When the doctor determines that the patient who has attended the Endocrinology and Nutrition Day Hospital needs to start glucose monitoring and goes to the nursing office, if he meets the inclusion criteria, he will be asked to participate in the study. After signing the informed consent, the control group (MGC) or intervention group (FSL2) will be randomised. The necessary therapeutic education for glucose monitoring will be carried out in parallel with the other necessary aspects of Diabetes Therapeutic Education.

Follow-up visits in both groups will take place 24-48 hours after the first visit, a week, 2 weeks, and 1, 2, and 3 months after the first visit. During visits, frequently according to usual clinical practice, by the nurse and/or doctor, therapeutic decisions will be made based on the monitoring system assigned to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM2.

  . Who have reached 18 years of age.
* Who are candidates to start glucose monitoring according to the usual clinical practice of the Endocrine Day Hospital of the Hospital de Sant Pau.
* That they are not using any glucose monitoring tool. These may be patients with debut diabetes, worsening control with high HbA1c levels, or starting treatment with glucocorticoids. Patients may have any of these conditions, or similar ones, as long as they meet the other inclusion criteria and none of the exclusion criteria. Similarly, no specifications are made for drug treatment prior to or initiated at the recruitment visit.

Exclusion Criteria:

* Pregnant or expecting to be during the duration of the study.
* Assessed by the healthcare professional responsible for proposing the study to them as more harmful than beneficial their inclusion in it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the treatment | 3 months
  Diabetes Treatment Satisfaction Questionnaire (DTSQ)

SECONDARY OUTCOMES:
Glucometrics | 3 months
  In each group, assess the change in blood glucose according to your monitoring method
The total number of visits | 3 months
  • The total number of visits (in person, by telephone and asynchronous telematics, if applicable).
Number of treatment | 3 months
  The number of treatment changes applied to the patient.
Duration of follow-up. | 3 months
  Duration of follow-up. A maximum follow-up of 3 months is expected in both groups. However, earlier completion is expected if the patient is discharged, requires hospital admission or an exclusion criterion is made before performing V7
HbA1c | Baseline and 3 months
  The hemoglobin A1c (HbA1c) test measures the amount of blood sugar (glucose) attached to your hemoglobin.
Perception of hiperglicemia | 3 months
  The value of questions 3 of the DTSQ and % of local problems as security variables.
Perception of hypoglicemia | 3 months
  The value of questions 2 of the DTSQ and % of local problems as security variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Natalia Mangas Fernandez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deshmukh H, Wilmot EG, Gregory R, Barnes D, Narendran P, Saunders S, Furlong N, Kamaruddin S, Banatwalla R, Herring R, Kilvert A, Patmore J, Walton C, Ryder REJ, Sathyapalan T. Effect of Flash Glucose Monitoring on Glycemic Control, Hypoglycemia, Diabetes-Related Distress, and Resource Utilization in the Association of British Clinical Diabetologists (ABCD) Nationwide Audit. Diabetes Care. 2020 Sep;43(9):2153-2160. doi: 10.2337/dc20-0738. Epub 2020 Jul 15. PMID 32669277
- [Background] American Diabetes Association Professional Practice Committee. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S83-S96. doi: 10.2337/dc22-S006. PMID 34964868
- [Background] Saisho Y. Use of Diabetes Treatment Satisfaction Questionnaire in Diabetes Care: Importance of Patient-Reported Outcomes. Int J Environ Res Public Health. 2018 May 9;15(5):947. doi: 10.3390/ijerph15050947. PMID 29747423
- [Background] Martens T, Beck RW, Bailey R, Ruedy KJ, Calhoun P, Peters AL, Pop-Busui R, Philis-Tsimikas A, Bao S, Umpierrez G, Davis G, Kruger D, Bhargava A, Young L, McGill JB, Aleppo G, Nguyen QT, Orozco I, Biggs W, Lucas KJ, Polonsky WH, Buse JB, Price D, Bergenstal RM; MOBILE Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Patients With Type 2 Diabetes Treated With Basal Insulin: A Randomized Clinical Trial. JAMA. 2021 Jun 8;325(22):2262-2272. doi: 10.1001/jama.2021.7444. PMID 34077499
- [Background] Diez-Fernandez A, Rodriguez-Huerta MD, Miron-Gonzalez R, Laredo-Aguilera JA, Martin-Espinosa NM. Flash Glucose Monitoring and Patient Satisfaction: A Meta-Review of Systematic Reviews. Int J Environ Res Public Health. 2021 Mar 18;18(6):3123. doi: 10.3390/ijerph18063123. PMID 33803558
- [Background] Fokkert M, van Dijk P, Edens M, Barents E, Mollema J, Slingerland R, Gans R, Bilo H. Improved well-being and decreased disease burden after 1-year use of flash glucose monitoring (FLARE-NL4). BMJ Open Diabetes Res Care. 2019 Dec 9;7(1):e000809. doi: 10.1136/bmjdrc-2019-000809. eCollection 2019. PMID 31875133
- [Background] Krakauer M, Botero JF, Lavalle-Gonzalez FJ, Proietti A, Barbieri DE. A review of flash glucose monitoring in type 2 diabetes. Diabetol Metab Syndr. 2021 Apr 9;13(1):42. doi: 10.1186/s13098-021-00654-3. PMID 33836819
- [Background] Bergenstal RM, Kerr MSD, Roberts GJ, Souto D, Nabutovsky Y, Hirsch IB. Flash CGM Is Associated With Reduced Diabetes Events and Hospitalizations in Insulin-Treated Type 2 Diabetes. J Endocr Soc. 2021 Feb 2;5(4):bvab013. doi: 10.1210/jendso/bvab013. eCollection 2021 Apr 1. PMID 33644623
- [Background] Evans M, Welsh Z, Ells S, Seibold A. The Impact of Flash Glucose Monitoring on Glycaemic Control as Measured by HbA1c: A Meta-analysis of Clinical Trials and Real-World Observational Studies. Diabetes Ther. 2020 Jan;11(1):83-95. doi: 10.1007/s13300-019-00720-0. Epub 2019 Oct 31. PMID 31673972
- [Background] Castellana M, Parisi C, Di Molfetta S, Di Gioia L, Natalicchio A, Perrini S, Cignarelli A, Laviola L, Giorgino F. Efficacy and safety of flash glucose monitoring in patients with type 1 and type 2 diabetes: a systematic review and meta-analysis. BMJ Open Diabetes Res Care. 2020 Jun;8(1):e001092. doi: 10.1136/bmjdrc-2019-001092. PMID 32487593
- [Background] Haak T, Hanaire H, Ajjan R, Hermanns N, Riveline JP, Rayman G. Flash Glucose-Sensing Technology as a Replacement for Blood Glucose Monitoring for the Management of Insulin-Treated Type 2 Diabetes: a Multicenter, Open-Label Randomized Controlled Trial. Diabetes Ther. 2017 Feb;8(1):55-73. doi: 10.1007/s13300-016-0223-6. Epub 2016 Dec 20. PMID 28000140
- [Background] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581